CLINICAL TRIAL: NCT02262325
Title: A Phase II Trial Combining Hypofractionated Radiation Boost With Conventionally-Fractionated Chemoradiation in Locally Advanced Non-small Cell Lung Cancer Not Suitable for Surgery
Brief Title: Hypofractionated Boost Before Chemoradiation for Patients With Stage II-III Non-small Cell Lung Cancer Unsuitable for Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Eric Miller, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14091; NCI-2014-01663 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-10-07; First posted 2014-10-13 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
Keywords: Non-small cell; Lung Cancer; Chemoradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; Etoposide; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (hypofractionated radiation boost, chemoradiation) (Experimental): Patients undergo hypofractionated radiation boost over 2 fractions (at least 40 hours apart) during week 1. Beginning week 2, patients receive cisplatin IV on days 8, 15, 36, and 43; and etoposide IV over 60 minutes on days 8-12 and 36-40. Patients also undergo standard 3-D conformal radiation therapy QD 5 days a week for a total of 30 fractions. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: hypofractionated radiation therapy; Drug: cisplatin; Drug: etoposide; Radiation: 3-dimensional conformal radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — Radiation boost in week 1 (days 1-5)
  Other Names: SBRT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving a hypofractionated boost to the primary tumor before standard chemotherapy and radiation therapy works in treating patients with stage II or III non-small cell lung cancer that cannot be removed by surgery. Advances in radiation oncology have allowed better radiation targeting which may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells. Giving more precise and targeted radiation before standard chemotherapy and radiation therapy may kill more tumor cells and prevent the cancer from coming back in the location in which it started.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the primary tumor control rate at 12 months.

SECONDARY OBJECTIVES:

I. To further establish safety and tolerability of this regimen. II. To estimate the rates of regional, distant control as well as progression-free survival and overall survival.

III. To evaluate the objective response rate (ORR) to this regimen. IV. To evaluate the response of tumors to stereotactic (high-dose) radiation using magnetic resonance tumor perfusion imaging modalities (magnetic resonance [MR]-dynamic contrast-enhanced [DCE]/perfusion weighted imaging [PWI], MR-diffusion, blood oxygenation level dependent [BOLD] sequences).

OUTLINE:

Patients will receive a hypofractionated boost to the primary tumor over 2 fractions (at least 40 hours apart) during week 1. Beginning week 2, patients receive cisplatin intravenously (IV) on days 8, 15, 36, and 43; and etoposide IV over 60 minutes on days 8-12 and 36-40. If carboplatin and paclitaxel is administered concurrently with radiotherapy, 2 cycles of carboplatin (AUC=6 mg/min/mL IV on day 1, 22) and paclitaxel (200 mg/m2 IV on day 1, 22) consolidation chemotherapy are required, to be administered starting 4-6 weeks after concurrent chemoradiation has ended. Each cycle is 21 days long. If cisplatin and etoposide is administered concurrently with radiotherapy, consolidation chemotherapy is not allowed. Patients also undergo standard conformal radiation therapy once daily (QD) 5 days a week for a total of 30 fractions. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0) =< grade 1 (except alopecia) at the time of enrollment
* Adequate baseline organ function obtained within 30 days of study registration
* Absolute neutrophil count >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine =< 1.5 ULN AND
* Calculated creatinine >= 50 mL/min (calculated by the Cockcroft-Gault formula) or
* 24-hour urine creatinine clearance >= 50 mL/min
* Non-small cell lung cancer (NSCLC), histologically and/or cytologically proven
* Clinical American Joint Committee on Cancer (AJCC) stage (7th edition) IIA-IIIB NSCLC (T1-4N1-3M0)
* Patients must be considered unresectable or medically-inoperable
* Patients must have primary tumor =< 6 cm as defined by CT largest axial dimension
* Within 60 days of registration: patients must have fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)-CT scan (or CT chest/abdomen/pelvis with IV contrast), and magnetic resonance imaging (MRI) brain with IV contrast (or CT scan of the brain with contrast); a non-contrast MRI scans of the chest/abdomen/pelvis or brain are permitted for workup if patient has allergy to CT contrast or renal insufficiency
* Within 30 days of registration: patients must have vital signs, history/physical examination, laboratory studies (complete blood count panel [CBCP] with differential, chemistries including liver function tests, creatinine clearance [CrCl] assessment, pregnancy test if needed within 14 days of registration)
* If a pleural effusion is present and visible on both CT scan AND chest x-ray, the investigator should exclude malignant disease by pleurocentesis to confirm cytologically-negative pleural fluid; if fluid is exudative or cytologically positive for tumor cells, patient is excluded
* Patients with effusions that are minimal (i.e. not visible on chest x-ray) and that are too small to safely tap are eligible.
* Life expectancy of at least 12 weeks in the opinion of investigator
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 30 days of registration
* Patients must have measurable primary tumor (undetectable NSCLC primary tumor is ineligible)
* Patients must be a minimum of 3 weeks from thoracotomy (if performed) and well-healed before starting treatment
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of registration; urine human gonadotropin (HCG) is an acceptable pregnancy assessment
* Nursing women may participate only if nursing is discontinued
* Women/men of reproductive potential must be counseled on contraception/abstinence while receiving the study treatment

Exclusion Criteria:

* Patients with contralateral hilar involvement (greater than 1.5 cm on short axis or positive on PET scan, or biopsy-proven)
* Documented or pathologically-proven metastatic disease
* Presence of nodules considered neoplastic in the same lobe or other ipsilateral lobe as the primary tumor (stage T3-4), unless the nodule can be encompassed in the stereotactic boost (gross tumor volume [GTV]boost) without exceeding a total GTVboost size of 6 cm as defined by CT largest axial dimension
* Presence of nodules considered neoplastic in contralateral lobes (M1a)
* Patients with history of pneumonectomy
* Prior cytotoxic chemotherapy or molecularly-targeted agents (e.g. erlotinib, crizotinib), unless > 2 years prior
* Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, or carcinoma in situ of the cervix; patients with a previous malignancy without evidence of disease for >= 3 years will be allowed to enter the trial
* History of active connective tissue disease (scleroderma) or idiopathic pulmonary fibrosis
* History of previous radiation therapy which would result in overlapping radiation fields
* Uncontrolled neuropathy grade 2 or greater, regardless of cause
* Subjects who are breast-feeding and plan to continue breast-feeding during therapy, or have a positive pregnancy test will be excluded from the study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Medical contraindication to MR imaging (e.g. pacemakers, metallic implants, aneurysm clips, known contrast allergy to Gadolinium contrast, pregnancy, nursing mothers, weight greater than 350 pounds) [first 10 patients]
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator; this could include severe, active co-morbidities such as:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last months
  * Transmural myocardial infarction within the last 6 months
  * Acquired immune deficiency syndrome (AIDS) based upon the current CDC definition; note, however, that HIV testing is not required for entry to protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved may be significantly immunosuppressive
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic insufficiency resulting in jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Miller, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Started | 21
Completed | 4
Not Completed | 17
Not completed — Death | 16
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Primary Tumor Control Rate, as Measured From the Time of Treatment Completion Until the First Documented Date of Local Failure
Description: Primary tumor control rate at 12 months, as well its 95% confidence interval, will be reported for all eligible subjects received treatment.
Time Frame: At 12 months following chemo/radiation therapy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants | 100

2. Secondary Outcome: Number of Adverse Events
Description: Number of all adverse events with special attention to grade 3-5 esophagitis, pneumonitis, and cardiac adverse events as defined by the National Cancer Institution Common Terminology Criteria for Adverse Events CTCAE version 5.0
Time Frame: Up to 30 days after completion of treatment, up to 5 years
Measure: Number; unit: Number of Events
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
Number of Events
  Abdominal Pain | 2
  Activated partial thromboplastin time prolonged | 1
  Acute kidney injury | 1
  Adrenal insufficiency | 1
  Alanine aminotransferase increased | 2
  Alopecia | 11
  Anemia | 14
  Anorexia | 7
  Aortic valve disease | 1
  Arthralgia | 1
  Aspartate aminotransferase increased | 3
  Bloating | 1
  Blood and lymphatic system disorders- Other, coagulation | 1
  Blurred vision | 1
  Bronchial infection | 1
  Bronchial obstruction | 1
  Bronchial stricture | 1
  Bruising- Lt rib area | 1
  Chest wall pain | 1
  Chills | 1
  Confusion | 1
  Constipation | 6
  Cough, intermittent | 4
  Cushingoid, face | 1
  Dehydration | 7
  Dermatitis Radiation (to upper back and skin darkening to the underside of right breast) | 15
  Diarrhea | 6
  Dizziness | 6
  Dysgeusia | 1
  Dyspepsia | 2
  Dysphagia | 14
  Dyspnea | 7
  Dyspnea and cough | 3
  Ear and labyrinth disorders- Other, Chronic otomastoiditis- bilateral | 1
  Epistaxis | 1
  Esophageal pain- odynophagia | 3
  Esophageal stenosis | 1
  Esophagitis | 14
  Fall | 1
  Fever (Max 100.8) | 2
  Fibrosis deep connective tissue | 1
  Flushing | 1
  Fracture- left rib | 1
  Gastritis | 1
  Gastroesophageal reflux disease (GERD) | 2
  Gastrointestinal disorders- Other- Perirectal abscess | 2
  Headache | 2
  Hematuria | 2
  Hiccups | 3
  Hoarseness | 1
  Hyperglycemia | 2
  Hyperkalemia | 1
  Hypernatremia | 1
  Hyperpigmentation- left chest (red discoloration) | 2
  Hypertension- intermittent | 3
  Hypoalbuminemia | 2
  Hypocalcemia (uncorrected- 8.3) | 2
  Hypokalemia (3.3) | 5
  Hypomagnesemia (1.5) | 4
  Hyponatremia | 2
  Hypophosphatemia | 1
  Hypotension- orthostatic | 1
  Hypothyroidism | 1
  Hypoxia | 1
  Infections and infestations- Other- Bacteremia | 2
  Infusion related reaction during Paclitaxel infusion | 2
  Infusion site reaction- right forearm- General disorders other | 2
  Insomnia | 1
  Localized edema- left chest wall | 1
  Lung infection-pneumonia | 5
  Lymphocyte Count Decreased | 19
  Mucosal infection- mouth thrush | 2
  Musculoskeletal and connective tissue disorder- Other, right paraspinal muscle spasm | 2
  Mucositis oral- mouth sore | 3
  Myalgia | 1
  Nasal congestion | 1
  Nausea | 10
  Nervous system disorders- Other, increased sense of smell, intermittent | 4
  Neutrophil count decreased | 9
  Non-cardiac chest pain | 4
  Pain in extremity- both hands due to arthritis | 2
  Pain- back | 2
  Pain-ribs | 1
  Palpitation | 1
  Paresthesia- both lower extremities | 1
  Pericardial effusion | 2
  Peripheral motor neuropathy | 2
  Peripheral sensory neuropathy | 4
  Platelet count decreased | 11
  Pleural effusion | 5
  Pleuritic pain, intermittent (Rt below breast) | 1
  Pneumonitis, radiation related | 8
  Productive cough | 7
  Proteinuria | 1
  Pruritis (back) | 1
  Pulmonary fibrosis | 9
  Rash- maculo-papular- back/chest | 3
  Respiratory failure | 1
  Respiratory, mediastinal and thoracic disorders- Other- COPD | 4
  Sebaceous cyst on the back | 3
  Sepsis | 1
  Sinus bradycardia | 1
  Sinus tachycardia | 2
  Skin infection- gluteal cleft | 2
  Sore throat | 3
  Syncope | 1
  Tachycardia- intermittent | 3
  Tinnitus- both ears | 2
  Tremor | 1
  Upper respiratory infection | 2
  Urinary Tract Infection- Pyelonephritis | 2
  Vomiting- intermittent | 9
  Weight gain | 1
  Weight loss | 7
  Wheezing | 6
  White blood cell count decreased | 17
  Fatigue | 11

3. Secondary Outcome: Tolerability Measured by the Number of Patients Who Discontinue Treatment
Description: The number of patients who discontinue treatment will be summarized.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
participants | 0

4. Secondary Outcome: Regional Control
Description: Regional control rate at 24 months will be reported for all eligible patients who received treatment.
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants | 81.6

5. Secondary Outcome: Distant Control
Description: Distant control rate at 24 months will be reported for all eligible patients who received treatment
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants | 70.3

6. Secondary Outcome: Disease-free Survival (DFS)
Description: Kaplan-Meier (K-M) analysis will be used to estimate DFS.
Time Frame: From date of treatment initiation to progression, assessed up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants | 46.1

7. Secondary Outcome: Overall Survival (OS)
Description: K-M analysis will be used to estimate OS.
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants | 50.3

8. Secondary Outcome: Objective Response Rate as Measured by Response Evaluation Criteria in Solid Tumors Criteria
Description: Objective response rate will be reported for all eligible patients who receive treatment.
Time Frame: At 3 months and 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 21
percentage of participants
  At 3 months | 72.7
  At 6 months | 80.0

9. Secondary Outcome: Changes in Tumor Perfusion Measured by MR-DCE/PWI Amp and Kep
Description: Changes in perfusion will be tested by comparing mean values pre- and post-hypofractionated boost radiation using a paired t-test. The following pharmacokinetic parameters will be used (parameters were derived using the modified Brix's model): Amp, Kep.
Time Frame: Baseline to the end of week 1
Population: The functional MRI substudies that measured changes in tumor perfusion were optional for participants. Eleven participants chose to participate in the substudies.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 11
percentage of change
  Changes in Kep | 2.9 (47)
  Changes in Amp | -6.8 (22.9)

10. Secondary Outcome: Changes in Tumor Perfusion Measured by MR-DCE/PWI Kpe and Kel
Description: Changes in perfusion will be tested by comparing mean values pre- and post-hypofractionated boost radiation using a paired t-test. The following pharmacokinetic parameters will be used (parameters were derived using the modified Brix's model): Kpe, Kel.
Time Frame: Baseline to the end of week 1
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 11
percentage of change
  Changes in Kpe | 5.1 [-11.1 to 24.6]
  Changes in Kel | -4.5 [-87.0 to 75.0]

11. Secondary Outcome: Changes in Diffusion Measured by MR-diffusion
Description: Changes in diffusion will be tested by comparing mean values of Apparent Diffusion Coefficient (ADC [× 10-3 mm2/s]) pre- and post-hypofractionated boost radiation using a paired t-test.
Time Frame: Baseline to the end of week 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 11
percentage of change | 23 (52.4)

12. Secondary Outcome: Changes in Hypoxia Measured by BOLD Sequences
Description: Changes in hypoxia will be tested by comparing mean values pre- and post-hypofractionated boost radiation using a paired t-test.
Time Frame: Baseline to the end of week 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
Number analyzed (Participants) | 11
percentage of change | -87.1 (144.7)

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Treatment (Hypofractionated Radiation Boost, Chemoradiation)
All-Cause Mortality (participants affected / at risk) | 16/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated Radiation Boost, Chemoradiation) (N=21)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Perirectal Abscess (Gastrointestinal disorders) | 1 (1)
Hypotenstion- orthostatic (Vascular disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Lung Infection - pneumonia (Infections and infestations) | 2 (2)
Hernia just superior to umbilicus (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonitis, radiation related (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event, Bilateral lower extremity deep vein thrombosis (Vascular disorders) | 1 (1)
Urinary tract infection - pyelonephritis (Infections and infestations) | 2 (2)
Atherosclerosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated Radiation Boost, Chemoradiation) (N=21)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction to an elastic bandage wrap (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 18 (18)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Aortic Valve Disease (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Coagulation (Blood and lymphatic system disorders) | 2 (2)
Blurred vision (Eye disorders) | 4 (4)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 4 (4)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (11)
Cough, intermittent (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Investigations) | 5 (5)
Cushingoid, face (Endocrine disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Depression (Psychiatric disorders) | 4 (4)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dizziness (Nervous system disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 14 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnea and cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Chronic otomastoiditis - bilateral (Ear and labyrinth disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Esophageal pain - odynophagia (Gastrointestinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 14 (14)
Vision Change (Eye disorders) | 2 (2)
Fall (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02262325/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02262325/ICF_001.pdf